#### **Information Sheet**

Study Title: Evaluation of an Interactive Computer-based Intervention to Safe Sex Practice for Female

**University Students: A Multicentred Randomized Controlled Trial** 

**Researcher:** Dr Janet Yuen Ha Wong **Institution:** The University of Hong Kong

#### Introduction

You are being invited to participate in an evaluation study from the University of Hong Kong. Please take time to read the information below and ask question whenever you find anything you do not understand, before deciding whether or not you wish to take part.

## 1. What is the purpose of the study?

The study is designed to evaluate the efficacy of an Interactive Computer-based Intervention (ICBI) to enhance safe sex practice among female university students.

### 2. Do I have to take part?

Your participation is entirely voluntary. Your choice of participation will not influence any of your relations to the University of Hong Kong. If you decide to participate, you are also free to withdraw any time without penalty.

# 3. What will happen to me if I take part?

You are going to administer a set of web-based questionnaires at the enrolment of the study. Then, you will be randomized to either intervention group or control group and have access to web-based sexual health information. The time spent on the web information will approximately be 30 minutes for intervention group and 10 minutes for control group. After the entry of study at 3-month and 6-month, you are going to administer a follow-up questionnaire online.

### 4. What are the risks of taking part?

There are no known risks of participating in this study.

## 5. What are the anticipated benefits of taking part?

Information from this study may benefit the development of more effective computerized sexual health intervention and you will be equipped with enhanced knowledge, attitude, norms, and self-efficacy of adopting safer sex practice.

## 6. Will my taking part in this study be kept confidential?

This study is anonymous and all the information will be kept confidential. You are only identified by participant identification number. If necessary, you have access to your personal data and the results of this study.

Under the Hong Kong law, the Personal Data (Privacy) Ordinance, Chapter 486, you can enjoy your personal information be kept confidential to protect the right. If you have any questions, please call the Privacy Commissioner's hotline (Tel: 2827 2827).

### 7. Who has reviewed the study?

Institutional Review Board of The University of Hong Kong / Hospital Authority Hong Kong West Cluster (HKU / HKW IRB) has reviewed the study. It is also one of the authorized parties to access your information related to the study for ethics review purpose.

# 8. Will I be charged for the study participation or receive any reward?

You will not be charged for the study participation. You will be offered \$100 vouchers after finishing the questionnaire at 3-month follow up and this \$100 voucher will be received upon the completion of questionnaire at 6-month follow up. Upon completion of both follow-up questionnaires, \$300 vouchers in total will be given.

# 9. Contact for further information

If you would like to know further details about the study, you are welcome to contact the principal researcher: Dr Janet Yuen Ha Wong of the School of Nursing, The University of Hong Kong (Tel: 3917 6641).

If you would like to know more about your right to participate in this study, please contact: Institutional Review Board of The University of Hong Kong / Hospital Authority Hong Kong West Cluster (HKU / HKW IRB) Secretary (Tel: 2255 4086).

#### 10. If I am willing to participate in this study, what do I have to do?

If you are willing to participate in this study, please sign an informed consent attached.

# **Informed Consent**

| <b>Study Title:</b> Evaluation of an Interactive Computer-based Intervention to Safe Sex Practice for Students: A Multicentred Randomized Controlled Trial <b>Researcher:</b> Dr Janet Yuen Ha Wong | or Female University |
|---|---|
| Participant Identification Number: | |
| <ol> <li>I confirm that I have read and understood the information sheet for the above study<br/>and have had the opportunity to ask questions. I will receive a copy of information<br/>sheet and informed consent form.</li> </ol> | Please check box "√" |
| 2. I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my services or legal rights being affected. | |
| 3. I understand that sections of any information given may be looked at by responsible individuals from the research team where it is relevant to my taking part in research. I give permission for these individuals to have access to my information and know all my information will be kept confidential. | |
| 4. I agree to take part in the above study. | |
| Name of Participant Signature Date | |
| Research Team | |
| Name of person taking consent/ Signature Date Researcher | |